CLINICAL TRIAL: NCT06449911
Title: Efficacy and Safety of High Intense Focused Ultrasound for Treating Middle and Lower Face and Submental Region Laxity
Brief Title: The Efficacy of Microfocused Ultrasound Technique in the Treatment of Facial Skin Laxity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0919
Record Dates: First submitted 2024-06-04; First posted 2024-06-10 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2023-12

CONDITIONS: Middle and Lower Face and Submental Region Skin Laxity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HIFU (Experimental): All participants will be treated using M4.5, level V, with 150 lines on the lower face and submental area; D4.5, level V, 10 Hz, with 4200 dots performed in 7 min on the lower face and the perioral and preauricular areas; M3.0, level V, with 150 lines on the lower face and submental area; D3.0, level V, 10 Hz, with 6000 dots performed in 10 min on the lower face, submental area, and middle face. The microfocused probes were uniformly set to a length of 25 mm with an interval of 1.5 mm. A total of 300 lines and 10,200 dots were performed for each half lower two-thirds of the face and submental area.
  Interventions: Procedure: HIFU

INTERVENTIONS:
Procedure: HIFU — 300 lines and 10,200 dots will be performed to each half lower two-thirds of the face and submental area of every participant.

SUMMARY:
This is a prospective study of 20 Chinese patients with lower facial laxity treated by High Intense focused ultrasound (HIFU). Response will be assessed via paired comparison of pretreatment and posttreatment photographs by two independent dermatologists, grading on a 5-point Subject Global Aesthetic Improvement Scale (SGAIS) for skin laxity. Quantitative analysis of submental lifting will also be performed. Patient's level of "sagging" and "volume loss", satisfaction and tolerance will be documented.

ELIGIBILITY:
Inclusion Criteria: healthy male or female, aged 30-60 years, seeking improved jawline definition, and/or reduction of submental skin laxity and were willing and able to provide informed consent.

Exclusion Criteria: Pregnancy or lactation, severe sun damage, excessive skin laxity on the lower face and neck, keloid scarring or open wounds in the treatment areas, severe or cystic facial acne, history of cosmetic treatments in the area to be treated (skin tightening procedure within the past year; injectable filler or botox within the past 6 months; ablative or nonablative resurfacing/rejuvenating laser treatment or light treatment within the past 6 months; dermabrasion or deep facial peels within the past 6 months), isotretinoin treatment within the past 6 months, and inability to understand the treatment protocol or to give informed consent.

Ages: 30 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
5-point Subject Global Aesthetic Improvement Scale (SGAIS) for skin laxity | 6 months after HIFU treatment
  0-worse, 1-0%-25% poor response, 2-25%-50% fair response, 3-50%-75% good response, 4-75%-100%-excellent response.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Dermatology, Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China